CLINICAL TRIAL: NCT07013188
Title: Characterising the Neuromuscular Function of Stroke Patients During Recovery
Brief Title: Characterising the Neuromuscular Function of Post Stroke Patients
Acronym: (cSTROKE)
Status: Recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Bethan Phillips, Professor, University of Nottingham
Other Study IDs: FMHS 188-0524
Record Dates: First submitted 2024-09-27; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-04

CONDITIONS: Stroke (CVA) or TIA
Keywords: Stroke; CVA; TIA; Neuromuscular
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Stroke patients: * Aged between 40-85 years
  * Willing and able to give informed consent for participation in the study
  * Had a confirmed stroke within the last 5 years
  * Self-reports persisting post-stroke loss of unilateral limb function
  Interventions: Other: Neuromuscular function

INTERVENTIONS:
Other: Neuromuscular function — Assessing their neuromuscular abilities using some functional and electromyography assessments

SUMMARY:
Strokes are a leading cause of death and disability in developed countries, with significant economic and social impacts. Defined by the WHO, strokes cause rapid and lasting disturbances in cerebral function. In the UK, strokes occur every five minutes, affecting 100,000 people annually and resulting in substantial physical impairments and financial costs. Although stroke-related deaths have decreased due to improved treatments and awareness, strokes remain a major cause of death and disability worldwide, especially in lower-income countries. Strokes typically cause unilateral deficits, leading to significant daily challenges and necessitating tailored rehabilitation strategies such as CIMT, FES, and VR Rehab. As the population ages, innovative neurorehabilitation approaches are essential to enhance functional recovery post-stroke. This pilot study aims to better understand the neuromuscular deficits caused by stroke to inform and improve future rehabilitation interventions, including the potential use of force accuracy training (FAT)

DETAILED DESCRIPTION:
In developed countries, strokes are the third most common cause of death and disability. Stroke is defined by the World Health Organization (WHO) as "rapidly developed clinical signs of focal (or global) disturbance of cerebral function, lasting more than 24 hours or leading to death, with no apparent cause other than of vascular origin. In 2013, the American Heart Association added the term "silent pathology" to the definition, which includes silent haemorrhage and infarctions of the brain, spinal cord, and retina. A transient ischemic attack (TIA) is considered a "warning stroke" because although it has similar symptoms to a stroke, the symptoms last for less than 24 hours. Furthermore, approximately 50% of strokes happen within 24 hours of a TIA.

The National Institute for Health and Care Excellence (NICE) estimates that in the UK a stroke occurs once every five minutes, and 100,000 people suffer from strokes annually. Further, over 1.3 million individuals in the UK have survived a stroke, with two-thirds of these survivors leaving the hospital with some physical impairment. There are 32,000 stroke-related fatalities annually in England alone, and stroke results in an annual expenditure in the region of £26-billion across the UK. In the previous 15 years, there has been a 49% decrease in the number of deaths caused by stroke in the UK despite an ageing population and that advancing age is a clear risk factor for stroke. This is likely due to advancements in both clinical treatment pathways and public awareness.

Despite this reduction in deaths, in terms of disability-adjusted life-years lost (DALY's), stroke is still the second-highest leading cause of death and is considered to be the third-leading cause of disability globally. In 2020, one in six cardiovascular disease-related deaths were caused by strokes. Global costs associated with stroke are projected to exceed 721 billion dollars (0.66 % of the global GDP). The burden (in terms of the absolute number of cases) grew dramatically from 1990 to 2019, with the bulk of worldwide stroke burden lying in lower and lower to middle-income countries (86.0% of fatalities and 89.0% of DALY's). This rise may be linked to a 70 % increase in incident of strokes, a 44 % increase in stroke-related mortality, a 102 % increase in general strokes, and a 143 % increase in prevalent strokes. Therefore, stroke is a disease of immense importance to the global population's health, with significant repercussions for individuals, the economy and society. In the past, it was believed that stroke primarily impacted wealthy nations. In contrast, the burden of stroke has fallen dramatically in many developed countries due to the use of evidence-based management techniques.

One hallmark of stroke is its tendency to cause unilateral deficits, affecting one side of the body. This can lead to weakness, paralysis, and sensory disturbances. These deficits pose significant challenges for daily activities and can have profound psychological and social impacts. Addressing these unique features is vital in rehabilitation, where tailored interventions can improve outcomes and quality of life for stroke survivors. Some of the current stroke rehabilitation strategies include Constraint-Induced Movement Therapy (CIMT), Task-Specific Training, Functional Electrical Stimulation (FES), Robot-Assisted Therapy, Virtual Reality (VR) Rehab, and Cognitive Rehabilitation. These approaches all aim to maximize recovery and improve functional outcomes post-stroke.

As the number of stroke survivors grows due to demographic shifts in our ageing societies, novel strategies for neurorehabilitation are required. Neural reorganisation is the most important driver of functional recovery after a stroke. An enhanced knowledge of the mechanisms that enable plasticity and recovery is required for the development of novel, neurobiologically informed techniques to promote functional recovery.

In sum, a better understanding of the neuromuscular deficits caused by stroke, which will be gained from this pilot study, will allow enhanced future design of rehabilitation interventions, and will inform the consideration of force accuracy training (FAT) as a potential intervention to improve the neuromuscular and physical function of stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* • Aged between 40-85 years

  * Willing and able to give informed consent for participation in the study
  * Had a confirmed stroke within the last 5 years
  * Self-reports persisting post-stroke loss of unilateral limb function

Exclusion Criteria:

* • Diagnosis of cognitive impairment/dementia

  * Current or recent (<2y) malignancy
  * Severe respiratory disease (e.g., uncontrolled asthma, COPD, pulmonary hypertension)
  * Active cardiovascular disease: Uncontrolled hypertension (BP>160/100mmHg); Recent (<12mo) cardiac event; Heart failure (Class III/IV); Significant arrhythmia; Unstable angina
  * Metabolic disease: Untreated hyper/hypoparathyroidism; Cushing's disease
  * Significant musculoskeletal disorders (based on clinical opinion)
  * Dialysis patients
  * Recent steroid treatment within 6 months or hormone replacement therapy
  * Mobility dependant (wheelchair dependency)

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-stroke survival
Sampling Method: Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Isometric dynamometry | During the single testing session (baseline) for the eligible stroke survivors who had a stroke within the past 5 years
  to determine maximum voluntary contraction (MVC) for upper and lower limb extension and flexion, including handgrip dynamometry (in Newton unit)
High-Density Surface electromyography (HDsEMG) and intramuscular electromyography (iEMG) of the muscles of the upper (bicep and tricep) and lower limbs (vastus lateralis and tibialis anterior) to determine muscle activation patterns | During the single testing session (baseline) for the eligible stroke survivors who had a stroke within the past 5 years
  Intramuscular electromyography (iEMG) and high-density sEMG (HD-sEMG) will be used to determine motor unit structure (size & number) and function (firing rate, firing complexity, neuromuscular junction transmission reliability). sEMG will also be used to determine muscle activation patterns and the largest compound muscle action potential (M-wave). This will be performed using skin electrodes (HDsEMG) and a small pin-type electrode (iEMG) inserted into the upper and lower limb muscles (measured in µVms).
Motor control assessments for the upper and lower limbs (i.e., force tracking tasks for knee and elbow extension). | During the single testing session (baseline) for the eligible stroke survivors who had a stroke within the past 5 years
  Participants will be requested to follow a force trace line on a monitor during extension and flexion movements. The intensity of this force will be relative to their individual capabilities (measured as CoV of force)
Balance tests | During the single testing session (baseline) for the eligible stroke survivors who had a stroke within the past 5 years
  Using a platform that can assess features such as Centre of Pressure (COP) and sway, participants will be asked to stand on both feet, and then on one foot with their eyes open and closed. Time to failure (i.e., need to place second foot on the floor and/or open eyes) will be recorded. A chair will be located behind participants for this assessment and a researcher will remain within touching distance. Participants will only be requested to complete the aspects of this assessment that they feel comfortable doing (measured in millimeter).

SECONDARY OUTCOMES:
The Grooved Pegboard Test to assess dexterity | During the single testing session (baseline) for the eligible stroke survivors who had a stroke within the past 5 years
  This simply involves participants placing small metal pegs into small holes in a specific order. This assessment is timed (in seconds).
The Trail Making Test (TMT) | During the single testing session (baseline) for the eligible stroke survivors who had a stroke within the past 5 years
  is a timed, neuropsychological test that involves visual scanning and working memory (measured in seconds).

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Derby Hospital branch, School of Medicine, University of Nottingham, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Access to personal (identifiable) information is limited only to research staff involved in the participation elements of this study, and to audit staff as detailed above.